CLINICAL TRIAL: NCT02072863
Title: Phase 1b/2, Multicenter, Open-label Study of Oprozomib, Melphalan, and Prednisone in Transplant Ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Oprozomib, Melphalan, and Prednisone in Transplant Ineligible Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPZ006; 2013-002125-27 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ONX 0912; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oprozomib with Melphalan and Prednisone (OMP) (Experimental): Subjects will receive oprozomib administered orally.
  The combination of oprozomib, melphalan, and prednisone (OMP) will be administered until progression of disease, unacceptable toxicity, discontinuation of study treatment for reasons other than progression or toxicity, or a maximum of 9 cycles (54 weeks), whichever occurs first.
  Interventions: Drug: Oprozomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Oprozomib — Study subjects will receive oprozomib administered orally.
Drug: Melphalan — Study subjects will receive melphalan 9 mg/m2.
Drug: Prednisone — Study subjects will receive prednisone 60 mg/m2.

SUMMARY:
The purpose of Phase 1b of the study is to determine the maximum tolerated dose (MTD) of oprozomib in combination with melphalan and prednisone (OMP).

The purpose of Phase 2 of the study is to estimate the overall response rate (ORR) and complete response rate (CRR) of the OMP combination.

ELIGIBILITY:
Key Inclusion Criteria:

1. Newly diagnosed symptomatic multiple myeloma patients who are transplant ineligible with measureable disease as indicated by one or more of the following:

   1. Serum M-protein ≥ 500 mg/dL
   2. Urine M-protein ≥ 200 mg/24 hour
   3. Serum Free Light Chain: Involved free light chain (FLC) level ≥ 10 mg/dL, provided serum FLC ratio is abnormal
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
3. Creatinine clearance (CrCl) ≥ 30 mL/min, either measured or calculated using the formula of Cockcroft and Gault [(140 - age) × mass (kg) / (72 × serum creatinine mg/dL)]. Multiply result by 0.85 if female.

Key Exclusion Criteria:

1. Any prior systemic antimyeloma therapy except oral steroids (dexamethasone up to a total dose of 160 mg or equivalent within 14 days prior to the first dose of study treatment is allowed). Use of topical or inhaled steroids is acceptable.
2. Congestive heart failure (New York Hearth Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to first dose
3. Known or suspected HIV, active Hepatitis A, B C or virus infection (Exception: Subjects with chronic or cleared HBV and HCV infection and stable liver function tests [bilirubin, AST] will be allowed).
4. Significant neuropathy (Grade 2 with pain or higher) at the time of first dose.
5. Plasma cell leukemia.
6. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
7. Known amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) - Phase 1b | 42 weeks
  MTD is defined as the highest dose at which a DLT is observed in less than 2 of 6 evaluable subjects occurring within the 4 weeks after the first dose of combination therapy.
Overall Response Rate (ORR) - Phase 2 | 39 months
  ORR defined as a best overall response of sCR, CR, VGPR, or PR according to the IMWG-URC.
Complete Response Rate (CRR) - Phase 2 | 39 months
  CRR defined as a best overall response of sCR or CR according to the IMWG-URC.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) - Phase 2 | Collected from signing of informed consent and throughout study until 30 days after the last dose of study treatment (up to 58 weeks)
  Adverse Events (AEs) and Serious Adverse Events (SAEs) graded according to the NCI-CTCAE (Version 4.03).
Population Pharmacokinetic (PK) parameters - apparent clearance and volume of distribution | 2 postdose time points in Cycle 1 Day 1, 1 predose and 2 postdose time points on Cycle 3 Day 1 and Cycle 5 Day 1
  Evaluate population pharmacokinetic (PK) parameter estimates of oprozomib and variability in these estimates when administered in combination with melphalan and prednisone using a sparse sampling strategy and population-based analysis methodology.
Duration of Response (DOR) | 39 months
  Duration of Response (DOR) is defined as the time from evidence of PR or better to disease progression or death due to any cause.
Progression-free Survival (PFS) | 39 months
  Progression-free survival is defined as the time from the first day of study treatment (Cycle 1 Day 1) to the earlier of disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- Department of Clinical Therapeutics, University of Athens, Athens, Attica, Greece
- Italy (5):
  - Ospedale Oncologico Regionale, Rionero in Vulture, Potenza
  - Azienda Ospedaliera Universitaria S Martino, Genova
  - AOU Maggiore della Carita, SCDU Heamatology, Novara
  - University of Rome, Rome
  - Hospital City of Health and Science of Turin, Hematology 1 Division, Turin
- Netherlands (2):
  - Vrijc Universiteit Medisch Centrum, Department of Hematology, Amsterdam
  - Erasmus MC, Department of Hematology, Rotterdam